CLINICAL TRIAL: NCT05862259
Title: A Multicenter, Multiomics, Non-interventional, Real-world Study of the Efficacy and Safety of Immune Checkpoint Inhibitors as First-line Therapy for Advanced Malignancies
Brief Title: A Real-world Study of the Efficacy and Safety of ICIs as First-line Therapy for Advanced Malignancies
Status: Recruiting | Type: Observational
Sponsor: Xinqiao Hospital of Chongqing (Other)
Responsible Party: Principal Investigator, Jianguo Sun, Deputy director of oncology department，clinical professor, Xinqiao Hospital of Chongqing
Other Study IDs: XQonc-021
Record Dates: First submitted 2023-05-08; First posted 2023-05-17 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Malignant Tumor; Immunotherapy; Artificial Intelligence
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, we collected the data of immunohistochemistry, gene detection, image, OS, PFS, Orr, and so on. Secondly, the database of immunotherapy for malignant tumor was established, and the predictive model was constructed to verify and establish the rationality and validity of the biomarkers and predictive system of immunotherapy

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent has been signed and, in the judgment of the investigator, the patient is able to comply with the study protocol and sign a written informed consent.
2. the advanced malignant tumors (solid tumors of the non-small-cell lung carcinoma, stomach, breast, urinary system, etc.) were diagnosed by histopathology.
3. the stage IV according to the eighth edition of IASLC.
4. PS 0-2, the expected survival > 3 months.
5. the age of 18-75 years.
6. no contraindication to treatment with immune checkpoint inhibitors.

Exclusion Criteria:

1. the patients' compliance was poor, which violated the rules of the trial;
2. the patients with severe dysfunction of vital organs (heart, liver and kidney) ;
3. the patients with other malignant tumors;
4. the researchers considered that the patients should not participate in other conditions of the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: receiving immunotherapy
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-08-10 (Actual); Primary Completion 2025-08-10 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | six months
  The time between randomization and the first occurrence of disease progression or death from any cause

SECONDARY OUTCOMES:
Overall survival | two years
  Time from randomization to death from any cause
Objective response rate | one years
  Proportion of patients whose tumors have shrunk to pre-defined volumes and who are able to maintain minimum time requirements
Immune-Related Adverse Events | two years
  In clinical trials of antineoplastic drugs/therapies, all levels of adverse drug reactions that are judged to be related to immune mechanisms,

OTHER OUTCOMES:
Indicators of cardiac injury | two years
  Including but not limited to troponin, BNP and cardiac magnetic resonance imaging

CONTACTS AND LOCATIONS:
Locations (1):
- the second affiliated hospital of Army medical university, Chongqing, Chongqing Municipality, China